CLINICAL TRIAL: NCT00000382
Title: Preventive Intervention for Maltreated Infants
Brief Title: Preventing Child Abuse in Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: R01MH054643 (NIH); R01MH054643 (NIH); DSIR CT-P
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Child Abuse
Keywords: Child Abuse; Female; Human; Infant; Male; Caregivers; Patient Education; Psychotherapy; Child Abuse -- *prevention & control
MeSH Terms: interventions — Child Protective Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Infant-Parent Psychotherapy
Behavioral: Child Protective Services
Behavioral: Psychoeducational Home Visitation
Behavioral: Parent Education

SUMMARY:
The purpose of this study is to compare 2 approaches (interventions) to prevent child-abuse (maltreatment) in infants: Psychoeducational Home Visitation (PHV) vs Infant-Parent Psychotherapy (IPP). Non-maltreated infants and their mothers are studied as a comparison group.

Twelve-month-old infants and their mothers are assigned randomly (like tossing a coin) to receive 1 of 3 types of intervention for 12 months: 1) Services normally available in the community when a family is reported for child maltreatment (Child Protective Services, CPS); 2) CPS involvement plus weekly PHV; 3) CPS involvement plus weekly IPP. Intervention will be provided until the infant's second birthday. All mother-infant pairs (including comparison non-maltreated infants and their mothers) will be assessed when the infant is 12, 18, 24, 36, and 48 months old. Assessments will look at the effectiveness of the intervention in preventing child maltreatment, improving parenting, and reducing future abuse. The study will last for 3 years.

Eligibility includes a mother and her 12-month-old child that has been abused by her (the mother) or the father. (Non-maltreated infants and their mothers also will be enrolled.)

DETAILED DESCRIPTION:
To evaluate the relative effectiveness of 2 theoretically-informed approaches to preventing the adverse sequelae of maltreatment in infants: Psychoeducational Home Visitation (PHV) and Infant-Parent Psychotherapy (IPP). Non-maltreated infants and their mothers serve as a comparison.

Maltreated infants and their mothers are randomly assigned to 1 of 3 types of intervention for 12 months: 1) Services routinely available in the community when a family is reported for child maltreatment (Child Protective Services, CPS); 2) CPS involvement plus weekly PHV; 3) CPS involvement plus weekly IPP. Intervention is provided until the infant's second birthday. All mother-infant dyads (including comparison non-maltreated infants and their mothers) participate in baseline assessments at the infant's age of 12 months. Subsequent assessments occur at 18, 24, 36, and 48 months of age. Assessments measure three major areas: 1) family-ecological variables; 2) maternal functioning and parenting; and 3) child functioning and stage-salient issues. CPS records are monitored annually across all groups to determine whether any reports of maltreatment have been filed.

ELIGIBILITY:
Inclusion Criteria:

-

Participants must have:

Infants that have been maltreated by their biological caregiver during their first year of life and who continue to reside with their maternal caregiver. (Non-maltreated infants and their mothers will also be enrolled.)

Ages: 12 Months to 12 Months | Sex: All
Age Groups: Child
Dates: Start 1998-07; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dante Cicchetti, PhD, Principal Investigator